CLINICAL TRIAL: NCT04006574
Title: Investigation the Effects of Core Stabilization Training on Gait, Balance, Muscle Strength, Functions, Fear of Movement and Quality of Life in Individuals With Developmental Hip Dysplasia
Brief Title: Developmental Hip Dysplasia and Physical Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Esra ATEŞ NUMANOĞLU, Research assistant, Ortopaedic Rehabilitation Department,Faculty of Physical Therapy and Rehabilitation, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-1357-18
Record Dates: First submitted 2019-06-27; First posted 2019-07-05 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Hip Dysplasia, Congenital
Keywords: Developmental Hip Dysplasia; Physiotherapy; Gait; Core Stabilization; Balance
MeSH Terms: conditions — Hip Dislocation, Congenital; Developmental Dysplasia of the Hip | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Single Blind Randomized Control Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- core stabilization training (Experimental): Patient with hip dysplasia aged between 20-60, non-operated
  Interventions: Other: Exercises
- traditional physiotherapy and core stabilization (Active Comparator): Patient with hip dysplasia aged between 20-60, non-operated
  Interventions: Other: Exercises

INTERVENTIONS:
Other: Exercises — Core stabilization
  Other Names: Traditional physiotherapy

SUMMARY:
Developmental Hip Displasia (DDH) can cause various degenerations or compensatory adaptations in the spine and knee joint, especially in the hip joint. As a result of adaptations and degeneration, these individuals may experience difficulty in walking and functional activities, lack of stabilization, decreased muscle strength and activation, and loss of balance at varying levels. This situation necessitates a holistic, multifaceted rehabilitation in individuals with hip dysplasia. There is no study in the literature that shows a specific physiotherapy and rehabilitation program applied to individuals with DDH. The aim of this study was to investigate the efficacy of classical physiotherapy method in patients with DDH and to compare the efficacy of classical physiotherapy and core stabilization exercise training in treatment.

DETAILED DESCRIPTION:
The study will be conducted in two groups. Individuals with DDH will be divided into two groups as conventional physiotherapy group and core stabilization group. It will be ensured that the distribution of the individuals in the groups in a randomized manner, with the disease stages of the two treatment groups being the same and the clinical characteristics are similar. The population of the study, individuals diagnosed with DDH by the orthopaedic surgeon, routinely directed to physiotherapy and rehabilitation, examined by the responsible investigator and who were referred to our clinic for the research, will be evaluated twice(before and after treatment) and will be treated for 3 times a week for 6 weeks. The study will consist of female individuals aged 20-60 who voluntarily agree to participate in the study (2 times evaluation and 18 times treatment). It is planned to involve at least 16 individuals. Individuals who meet the criteria for inclusion in the study and volunteers will be included in the study by signing the Informed Voluntary Consent Form. In Hacettepe University, Department of Physiotherapy and Rehabilitation, pain severity of subjects with DDH will be evaluated with Digital Analogue Scale (SAS) and algometer, joint range of motion with goniometer, muscle strength with digital dynamometer, walking with GaitRite device, balance with Bertec device and hip functions, kineyophobia, questionnaires will be given to evaluate quality of life and mood. After the first evaluation, individuals will be treated 3 times a week for 6 weeks and then the first evaluations will be done again. The data obtained before and after treatment will be compared between the two treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* age between 20-60 years old
* non-operated (total hip arthroplasty)

Exclusion Criteria:

* neurological disease
* cognitive problems

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — age between 20-60 years old, non-operated (total hip arthroplasty)
Enrollment: 16 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2020-01-16 (Actual)

PRIMARY OUTCOMES:
Hip Muscle Strength ( muscle isometric strength in Newton) | 6 weeks
  Muscle Strength will be evaluated by hand held dynamometer

SECONDARY OUTCOMES:
Hip Function | 6 weeks
  Hip Function will be evaluated with scale Harris Hip Score
Hip Pain | 6 weeks
  Pain will be evaluated with Digital Analog Scale in numbers 0-10

CONTACTS AND LOCATIONS:
Overall Officials: Esra ATEŞ NUMANOĞLU, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)